CLINICAL TRIAL: NCT00111189
Title: A Randomized Double-blind Placebo-controlled Parallel Group Study Evaluating Paliperidone Palmitate in the Prevention of Recurrence in Patients With Schizophrenia. Placebo Consists of 20% Intralipid (200 mg/mL) Injectable Emulsion.
Brief Title: A Study of the Efficacy (Effectiveness) of Paliperidone Palmitate in the Prevention of Recurrence of the Symptoms of Schizophrenia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CR004198; R092670PSY3001
Record Dates: First submitted 2005-05-17; First posted 2005-05-18 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone palmitate; R092670; antipsychotic; recurrence prevention
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): Paliperidone Palmitate 25, 50, 75 or 100 mg eq every 4 wk for up to 24 mo
  Interventions: Drug: Paliperidone Palmitate
- 002 (Placebo Comparator): Placebo Placebo every 4 wk up to 24 mo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo every 4 wk up to 24 mo
  Arms: 002
Drug: Paliperidone Palmitate — 25, 50, 75 or 100 mg eq every 4 wk for up to 24 mo
  Arms: 001

SUMMARY:
The purpose of this study is to evaluate the efficacy of paliperidone palmitate compared with placebo in the prevention of recurrence of the symptoms of schizophrenia and to assess the safety and tolerability of paliperidone palmitate in patients with stable and symptomatic schizophrenia. The placebo used in this study was a nutritional substance known as 20% Intralipid emulsion given to patients requiring intravenous feedings.

DETAILED DESCRIPTION:
Many patients with schizophrenia have difficulty adhering to a daily oral treatment regimen. Long-acting injectable formulations, such as long-acting injectable paliperidone palmitate, may provide therapeutic plasma concentrations over several weeks, thereby eliminating the need for daily oral medication and making compliance easier. This study is a randomized (patients will be assigned to different treatment groups based solely on chance), double-blind (neither the patient nor the physician will know if placebo or drug is being given and at what dose), placebo-controlled, parallel-group, multicenter study followed by an open-label extension period in patients with schizophrenia. The study is designed to evaluate the efficacy of paliperidone palmitate (a long-acting injectable formulation) in delaying the time to and decreasing the rate of recurrence compared with placebo in patients with schizophrenia. The study will consist of 5 periods: an up to 7-day screening/washout/tolerability period, a 9-week open-label transition period, a 24-week open-label maintenance period, a randomized, variable-length double-blind, placebo-controlled recurrence prevention period, and an up to 52-week open-label extension period. Patients will have intramuscular (i.m.) study drug injections and efficacy and safety evaluations performed every 4 weeks throughout the study. Efficacy will be evaluated during the study using a recurrence assessment, the Positive and Negative Symptom Scale for Schizophrenia (PANSS), the Clinical Global Impression - Severity (CGI-S) scale, and the Personal and Social Performance (PSP) scale. Safety will be assessed throughout the study by monitoring adverse events; use of extrapyramidal symptoms (EPS) rating scales (Abnormal Involuntary Movement Scale [AIMS], Barnes Akathisia Rating Scale [BARS], Simpson Angus Scale [SAS]); clinical laboratory testing; vital signs (temperature, blood pressure, and heart rate) measurements; electrocardiograms (ECGs); and physical examinations. Additionally, the patients will assess the tolerability of the injections by evaluating the pain of the injection and the pain at the injection sites. Tolerability test: 3 mg/day of oral ER OROS paliperidone for 4 days. Transition (9 wks): 50 mg eq. paliperidone palmitate i.m. dose on Day 1, then i.m. injections (25, 50, or 100 mg eq.) once every 4 wks (q4wk). Maintenance (24-wks): paliperidone palmitate i.m. injections (25, 50, or 100 mg eq.) q4wk. Recurrence Prevention: paliperidone palmitate i.m. injections (25, 50, or 100 mg eq. or placebo) q4wk. Open-label paliperidone palmitate (25, 50, 75, or 100 mg eq.) q4wk for 12 dosing periods.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the diagnostic criteria for schizophrenia according to DSM-IV-TM for at least 1 year before screening
* have a PANSS score of <120
* have a body mass index (BMI) >/=15.0 kilogram (kg)/meter (m)2
* and have resided at the same address for at least 30 days

Exclusion Criteria:

* Patients unable to provide their own consent
* have been involuntarily committed to psychiatric hospitalization
* have primary, active DSM-IV-TM diagnosis other than schizophrenia
* who have a DSM-IV-TM diagnosis of active substance dependence within 3 months before screening (nicotine and caffeine are not exclusionary)
* have a history of treatment resistance as defined by failure to respond to 2 adequate trials (minimum of 4 weeks at a therapeutic dose) of different antipsychotic medications
* have a history of any severe preexisting gastrointestinal narrowing or inability to swallow the medication whole with water
* have a history of neuroleptic malignant syndrome (NMS)
* are at significant risk of suicidal or violent behavior
* current presence of any significant or unstable medication condition
* treatment with any protocol disallowed therapies
* clinically significant result from screening laboratory or ECG.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2005-02; Primary Completion 2007-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The primary efficacy criteria for this study is the time from randomization to the first recurrence event during the double-blind recurrence prevention period | After 68 relapse events

SECONDARY OUTCOMES:
Changes from randomization to the end of the recurrence prevention period in PANSS (total and subscales), CGI-S, and PSP. Incidence of adverse events, labs and ECGs throughout study. | After 68 relapse events

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (55):
- United States (18):
  - Little Rock, Arkansas
  - Cerritos, California
  - Santa Ana, California
  - Hialeah, Florida
  - Chicago, Illinois
  - Granite City, Illinois
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
  - Flowood, Mississippi
  - St Louis, Missouri
  - Clementon, New Jersey
  - Cedarhurst, New York
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Conroe, Texas
  - DeSoto, Texas
  - Irving, Texas
  - San Antonio, Texas
- Costa Rica, Costa Rica
- Mexico (3):
  - Mexico City
  - Mérida
  - Monterrey
- Romania (6):
  - Bucharest
  - Cluj-Napoca
  - Iași
  - Sibiu
  - Tg Mures
  - Timișoara
- Russia (6):
  - Arkhangelsk
  - Moscow
  - Moscow Russia
  - Saint Petersburg
  - Samara
  - Yaroslavl
- South Africa (4):
  - Cape Town
  - Centurion Gauteng
  - Florida Johannesburg Gauteng
  - Johannesburg
- South Korea (4):
  - Gwangju
  - Inchun
  - Pusan
  - Seoul
- Taiwan (4):
  - Changhua
  - Kaohsiung City
  - Tainan
  - Taoyuan District
- Ukraine (9):
  - Dnipro
  - Hlevakha
  - Kharkiv
  - Kiev
  - Kyiv
  - Lviv
  - Odesa
  - Simferopol
  - Vinnitsa

REFERENCES:
- [Derived] Ceraso A, Lin JJ, Schneider-Thoma J, Siafis S, Tardy M, Komossa K, Heres S, Kissling W, Davis JM, Leucht S. Maintenance treatment with antipsychotic drugs for schizophrenia. Cochrane Database Syst Rev. 2020 Aug 11;8(8):CD008016. doi: 10.1002/14651858.CD008016.pub3. PMID 32840872
- [Derived] Mathews M, Gopal S, Singh A, Nuamah I, Pungor K, Tan W, Soares B, Kim E, Savitz AJ. Comparison of Relapse Prevention with 3 Different Paliperidone Formulations in Patients with Schizophrenia Continuing versus Discontinuing Active Antipsychotic Treatment: A Post-Hoc Analysis of 3 Similarly Designed Randomized Studies. Neuropsychiatr Dis Treat. 2020 Jun 19;16:1533-1542. doi: 10.2147/NDT.S221242. eCollection 2020. PMID 32606705
- [Derived] Emsley R, Nuamah I, Gopal S, Hough D, Fleischhacker WW. Relapse After Antipsychotic Discontinuation in Schizophrenia as a Withdrawal Phenomenon vs Illness Recurrence: A Post Hoc Analysis of a Randomized Placebo-Controlled Study. J Clin Psychiatry. 2018 Jun 19;79(4):17m11874. doi: 10.4088/JCP.17m11874. PMID 29924507
- [Derived] Weiden PJ, Kim E, Bermak J, Turkoz I, Gopal S, Berwaerts J. Does Half-Life Matter After Antipsychotic Discontinuation? A Relapse Comparison in Schizophrenia With 3 Different Formulations of Paliperidone. J Clin Psychiatry. 2017 Jul;78(7):e813-e820. doi: 10.4088/JCP.16m11308. PMID 28640988
- [Derived] Kozma CM, Slaton T, Dirani R, Fastenau J, Gopal S, Hough D. Changes in schizophrenia-related hospitalization and ER use among patients receiving paliperidone palmitate: results from a clinical trial with a 52-week open-label extension (OLE). Curr Med Res Opin. 2011 Aug;27(8):1603-11. doi: 10.1185/03007995.2011.595000. Epub 2011 Jun 22. PMID 21696265
- [Derived] Hough D, Gopal S, Vijapurkar U, Lim P, Morozova M, Eerdekens M. Paliperidone palmitate maintenance treatment in delaying the time-to-relapse in patients with schizophrenia: a randomized, double-blind, placebo-controlled study. Schizophr Res. 2010 Feb;116(2-3):107-17. doi: 10.1016/j.schres.2009.10.026. Epub 2009 Dec 2. PMID 19959339
- See also: A study of the efficacy of paliperidone palmitate in the prevention of recurrence of the symptoms of schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=564&filename=CR004198_CSR.pdf